CLINICAL TRIAL: NCT01848743
Title: Tenofovir Versus Lamivudine for Patients of Chronic Hepatitis B With Severe Acute Exacerbation
Acronym: HBSAE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Wei-Lun Tsai, Attending physician, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gilead IN-US-174- 0190
Record Dates: First submitted 2013-04-24; First posted 2013-05-07 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Chronic HBV With Severe Exacerbation
Keywords: tenofovir, lamivudine, hepatitis B, acute exacerbation
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir (Active Comparator): All enrolled patients are randomized to tenofovir arm who receives tenofovir 300 mg qd for 36 months
  Interventions: Drug: Tenofovir
- lamivudine (Placebo Comparator): All enrolled patients are randomized to lamivudine arm who received lamivudine 100 mg qd for 6 months, followed by tenofovir for another 30 months.
  Interventions: Drug: lamivudine

INTERVENTIONS:
Drug: Tenofovir
  Other Names: viread
  Arms: Tenofovir
Drug: lamivudine
  Other Names: zeffix
  Arms: lamivudine

SUMMARY:
In Taiwan, 15% of general population had hepatitis B virus (HBV) infection, HBV is the leading cause of liver cirrhosis and hepatocellular carcinoma in Taiwan. After entering immune clearance, 10-30% of patients of chronic HBV develop acute exacerbation (AE) , some are mild but some developed hepatic decompensation or even death.

Previous study found that early use of lamivudine before bilirubin level is above 20 mg/dl can improve survival in chornic HBV with severe AE. From the study from Hongkong, lamivudine was found to have better survival than entecavir in chronic HBV with severe AE. Recent study from India found that tenofovir is able to improve survival in chronic HBV with severe AE. The aim of this study is to compare the effect of lamivudine and tenofovir for chronic HBV with severe AE.

The study aims to enroll 120 patients with chronic HBV defined as persistence of HBsAg for more than 6 months. Severe AE was defined as ALT > 400 U/L, prolongation of prothrombin time > 3 seconds, bilirubin > 2 mg/dl. Patients with hepatitis A, C, D or HIV infection, drug or alcoholic liver disease, hepatocellular carcinoma, under immuno-suppressive agents use, or previous use of anti-HBV agents are excluded. All enrolled patients are randomized into group A who received tenofovir 300 mg qd for 3 years and group B who received lamivuidne 100 mg qd for 6 months, followed by tenofovir 300mg qd for 30 months. Mortality rate and virological, biochemical and serological response were evaluated at 1,2,4,48,96 and 144 weeks. The values are expressed as mean + SD. Categorical variables were analyzed with Chi-square test or Fisher's exact test as appropriate and continuous variables were analyzed by Mann-Whitney test. Logistic regression test was applied to analyze the independent association of various variables with outcome. A p value < 0.05 was regarded as significant.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg (+) > 6 months
* ALT > 5X ULN
* Prolongation of prothrombin time > 3 seconds and bilirubin level > 2 mg/dl
* 20-75 years old

Exclusion Criteria:

* HAV, HCV, HDV and HIV co-infection
* Concurrent hepatocellular carcinoma
* Drug, metabolic or alcohol as cause of hepatitis
* Anti-viral treatment in recent 6 mnths
* Pregnant woman

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
6 months survival | 6 months after treatment begins
  6 months survival after treatment begins

SECONDARY OUTCOMES:
rapid virological response | 1,2 and 4 weeks after treatment
  Evaluate the relationship of rapid virological response ( at 1,2 and 4 weeks) and survival
HBeAg seroconversion and virological response 1, 2, and 3 years after treatment | 1,2 and 3 years after treatment
  To evaluate the rate of HBeAg seroconversion and virological response 1, 2, and 3 years after treatment in the two arms
Safety profile | during and 6 months after treatment
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Veterans General Hospigal, Kaohsiung, Taiwan
  - Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan

REFERENCES:
- [Derived] Lu CM, Cheng JS, Sun WC, Chen WC, Tsay FW, Wang HM, Tsai TJ, Kao SS, Li YD, Li YR, Lin HS, Yin CH, Tsai WL. Randomized Controlled Study of Tenofovir versus Lamivudine Followed by Tenofovir in Severe Exacerbation of Hepatitis B. Antimicrob Agents Chemother. 2022 Feb 15;66(2):e0166421. doi: 10.1128/AAC.01664-21. Epub 2021 Nov 22. PMID 34807763